CLINICAL TRIAL: NCT04792099
Title: CPAP Or Nasal Cannula Oxygen for Preterm Infants: A Randomized Controlled Trial
Acronym: COCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Siamak Yazdi, Principal Investigator, Neonatology Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo ZY 2021
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Infant, Newborn, Disease; Hypoxia; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Disease; Hypoxia; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia | interventions — Continuous Positive Airway Pressure; Cannula

STUDY DESIGN:
Intervention Model Description: 1:1 parallel allocation of infants to CPAP or NC oxygen using randomization with stratified permuted block design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous positive airway pressure (Experimental): Continuous positive airway pressure (CPAP) with blended oxygen delivered by binasal prongs or nasal mask.
  Interventions: Procedure: Continuous positive airway pressure
- Nasal Cannula (Active Comparator): Blended oxygen delivered by nasal cannula (NC).
  Interventions: Procedure: Nasal Cannula

INTERVENTIONS:
Procedure: Continuous positive airway pressure — After study entry, CPAP will be provided via mask or binasal prongs in order to have a relatively uniform CPAP delivery system among infants in the treatment group. Bubble CPAP will be preferred over other modes of CPAP delivery. A PEEP of 5 will be used for uniformity.
  Other Names: CPAP
  Arms: Continuous positive airway pressure
Procedure: Nasal Cannula — After study entry, flow will be set to 0.5 L/kg with 1L maximum while on NC during the study period to reduce the risk of inadvertent PEEP with higher flows. Initial FiO2 can be titrated to achieve target saturations, and may be increased up to 100% while on NC.
  Other Names: NC
  Arms: Nasal Cannula

SUMMARY:
The purpose of this study is to determine if in preterm infants < 34 weeks' gestation at birth receiving respiratory support with continuous positive airway pressure (CPAP) or nasal cannula (NC), CPAP compared with NC will decrease the number of episodes with oxygen saturations less than 85% of ≥10 seconds in a 24-hour randomized controlled trial. This will be a randomized controlled trial with a 1:1 parallel allocation of infants to CPAP or NC oxygen using stratified permuted block design.

DETAILED DESCRIPTION:
We hope to determine whether in preterm infants < 34 weeks' gestation at birth receiving respiratory support with continuous positive airway pressure (CPAP) or nasal cannula (NC), CPAP compared with NC will decrease the number of episodes with oxygen saturations less than 85% of ≥10 seconds in a 24-hour randomized controlled trial.

This study will include preterm infants < 34 weeks' gestation on respiratory support via CPAP with a PEEP ≤ 5 and FiO2 ≤ 30%. There will be two randomization strata [≥ 22+0/7 to ≤ 27+0/7 weeks, and ≥ 27+1/7 to ≤ 33+6/7 weeks. The purpose of stratification is to ensure an appropriate distribution of risk between study arms. This study will not be powered to detect outcome differences within or between strata.

Following informed consent, randomization, stratified by gestational age at delivery, will be performed using sequentially numbered sealed opaque envelopes. Each envelope will indicate either Treatment group (CPAP group) or Control group (NC group). The envelope will only be opened after informed consent has been obtained and just before starting the study on each infant.

This will be a single center randomized controlled trial with a 1:1 parallel allocation of infants to CPAP or NC oxygen using stratified permuted block design. 15-30 minutes will be provided as a washout period at the beginning of the intervention, followed by 24 hours on the intervention. Infants enrolled must meet CPAP stability criteria that are based on prior randomized clinical trials of weaning from CPAP to NC.

All infants enrolled in the study will have routine monitoring, uniform target saturation ranges of 91-95% with alarm limits set at 88-95%, and standard care for the duration of the study. The high alarm limit will be increased to 100% if an infant is weaned to 21% FiO2. Supplemental FiO2 will be titrated per unit routine to achieve goal target saturations. Pulse oximetry recordings will be downloaded using ixTrend (iexcellence, Wildau, Germany) software to a secure computer system or via Bedmaster software for later data analysis. The target oxygen saturations (91 to 95%) are based on data from the meta-analysis of randomized controlled trials of oxygen saturation targets which included data on 4911 infants from the SUPPORT, COT, and BOOST II trials.

Primary and secondary outcomes are described below. Other safety outcomes include recordings of episodes of bradycardia and circumstances surrounding the event. Pulse oximetry recordings will be downloaded using ixTrend software to a secure computer system for later data analysis. Abdominal and cerebral NIRS will also be performed with subsequent data analysis..

ELIGIBILITY:
Inclusion Criteria:

* Infants must be currently utilizing CPAP (without a rate) with a PEEP ≤ 5 and FiO2 ≤ 30%
* Infants must meet CPAP stability criteria as follow:
* If previously intubated, must be extubated ≥ 72 hours
* < 3 self-resolving apneas (≤ 20 s) and/or bradycardia (< 100 bpm) in any hour over previous 6 hours)
* Gestational age < 34 weeks' gestation at birth
* Informed consent by parents/legal guardians

Exclusion Criteria:

* presence of a major malformation
* a neuromuscular condition that affects respiration
* a terminal illness or decision to withhold or limit support
* currently being treated for sepsis
* enrollment in a competing trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
The number of episodes with oxygen saturations less than 85% for ≥ 10 seconds | 24 hours of intervention

SECONDARY OUTCOMES:
The coefficient of variability of oxygen saturations (relative standard deviation) | 24 hours of intervention
  The coefficient of variation is a standardized measure of dispersion of a frequency distribution defined as the ratio of the standard deviation to the mean. It will be used in this study to assess the stability of oxygen saturations.
The proportion of time with oxygen saturations > 95 % among infants requiring supplemental oxygen | 24 hours of intervention
The proportion of time spent outside oxygen saturation target ranges (91-95%) among infants requiring supplemental oxygen | 24 hours of intervention
The proportion of time with oxygen saturations less than 85% | 24 hours of intervention
The median supplemental oxygen concentration | 24 hours of intervention
The median transcutaneous carbon dioxide value | 24 hours of intervention
The number of episodes (≥ 10 seconds) with oxygen saturations less than 80 % | 24 hours of intervention
The number of recorded episodes (≥ 10 seconds) of bradycardia < 100/min | 24 hours of intervention
The median cNIRS value | 24 hours of intervention
  Median cerebral near-infrared spectroscopy value during the 24 hour intervention period
The median aNIRS value | 24 hours of intervention
  Median abdominal near-infrared spectroscopy value during the 24 hour intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yazdi S, Carlo WA, Nakhmani A, Boateng EO, Aban I, Ambalavanan N, Travers CP. Extended CPAP or low-flow nasal cannula for intermittent hypoxaemia in preterm infants: a 24-hour randomised clinical trial. Arch Dis Child Fetal Neonatal Ed. 2024 Aug 16;109(5):557-561. doi: 10.1136/archdischild-2023-326605. PMID 38365446